CLINICAL TRIAL: NCT05700175
Title: Transcriptomic Study of Adult Population With Marfan Syndrome
Acronym: MaRfaNomicA
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Fabio Martelli, Dr, PhD, Molecular Cardiology Laboratory Director, IRCCS Policlinico S. Donato
Other Study IDs: MaRfaNomicA
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Marfan Syndrome; Marfan's Syndrome With Cardiovascular Manifestations
Keywords: Thoracic aortic aneurysm
MeSH Terms: conditions — Marfan Syndrome; Aortic Aneurysm, Thoracic | interventions — Epigenesis, Genetic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood aortic aneurysmal tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Transcriptomic, epigenetic and proteomic analysis — Next-generation sequencing will be used to identify differences in expression of circulating transcripts (protein-coding and not) in patients affected by Marfan Syndrome (MFS), subdivided based on the presence or absence of thoracic aortic aneurysms (TAA) and indication of TAA-surgery (TAA_MFS_signature).
  The obtained TAA_MFS_signature will be correlated to fundamental biological parameters by analysing:
  Blood-levels of cytokines and chemokines relevant for inflammation. Transcriptomic and epigenetic (Cytosine methylation) changes in aortic aneurysms tissue by Next-generation sequencing.
  Progression of biomarkers in surgical-patients before and at 6 and 12 months after surgery.

SUMMARY:
This project is designed to discover circulating biomarkers for aortic aneurysms in adults affected by Marfan Syndrome (MFS). The first aim is to identify circulating transcripts, protein-coding (mRNA) and not (ncRNAs), which show differential expression between three groups of adult patients affected by MFS, based on: presence or absence of thoracic aortic aneurysms (TAA) and indication of TAA-surgery. This obtained TAA_MFS_signature will then be correlated to fundamental biological parameters, like cytokines and chemokines relevant during inflammation and transcriptomic as well as epigenetics changes in aortic aneurysm tissue. Furthermore, the association of TAA_MFS_signature to genetic, clinical and instrumental parameters at present used for diagnosis and treatment, will be evaluated.

DETAILED DESCRIPTION:
The investigators will collect peripheral blood and aortic aneurysm tissues specimens from consenting subjects. For all three groups of MFS patients, total RNA will be isolated from peripheral whole blood, plasma and peripheral blood mononuclear cell (PBMC) and processed for transcriptomic analyses by RNAseq. Plasma will be used to determine cytokine and chemokine levels, using a luminex panel designed for inflammation biomarkers (serum proteomics). For all patients undergoing surgery, tissue specimens will be used for transcriptomic and epigenetic analysis, histological sections and serum proteomics.

ELIGIBILITY:
Inclusion Criteria:

General criteria:

* Clinically and genetically determined Marfan syndrome (according to the revised Ghent-criteria 2010)
* Signed informed consent
* Patient receiving regular pharmacological prophylaxis or newly diagnosed patients

Population without thoracic aortic aneurysms (TAA) Patients with clinically and genetically determined Marfan syndrome, presenting thoracic aortic diameters within established normal limits (mm and base Z-score).

Population with TAA "stable dimensions" Patients with clinically and genetically determined Marfan syndrome, presenting stable values for dimension / Z-score of the aortic root during the 12 months preceding the enrolment.

Population with TAA with surgery indication:

* Patients with clinically and genetically determined Marfan syndrome, presenting indication for surgical correctional according to the relevant International guidelines
* Trend of uncontrolled increase of aortic diameter compared to previous measurements
* Aortic ectasia associated to a clinically significant valve dysfunction
* Evaluation of cut-off for surgical intervention dependant also on familial dissection

Exclusion Criteria:

* Patients with chronic or acute inflammation states, like: chronic liver disease, chronic renal insufficiency (creatinine > 1.5 mg/dl) and diseases affecting the thyroid apparatus.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the IRCCS Policlinico San Donato.
Sampling Method: Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Transcriptomic Signature in adult patients suffering of affected by Marfan syndrome | year 1-5
  Identification of differences in transcript-expression between Marfan patients with or without thoracic aortic aneurysms (TAA) and with indication of TAA-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Martelli, Dr, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- Irccs Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No